CLINICAL TRIAL: NCT07384533
Title: Perioperative Recovery Outcomes of a Spontaneous Breathing-Preserving Strategy in Salvage Lung Transplantation: A Prospective Multicenter Single-Arm Clinical Study
Brief Title: Perioperative Recovery Outcomes of a Spontaneous Breathing-Preserving Strategy in Salvage Lung Transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Chief Physician and Professor of Thoracic Surgery, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BREATH-Rescue
Record Dates: First submitted 2026-01-21; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: End-stage Lung Disease
Keywords: Lung transplantation; Enhanced Recovery After Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tubeless LTx Group (Experimental): All participants receive lung transplantation under a standardized spontaneous-breathing-preserving ("tubeless") pathway. After anesthesia induction, a supraglottic airway (laryngeal mask airway) is used when feasible with regional nerve blocks and multimodal sedation/analgesia to control pain and cough while maintaining spontaneous breathing. Muscle relaxants are minimized; ventilatory assistance is provided only as needed with low airway pressures. Postoperatively, patients are managed in the intensive care unit with spontaneous breathing and protocol-guided noninvasive respiratory support. Conversion to endotracheal intubation, invasive mechanical ventilation, and/or extracorporeal membrane oxygenation is allowed if predefined safety criteria are met.
  Interventions: Procedure: Lung transplantation that preserves spontaneous breathing function

INTERVENTIONS:
Procedure: Lung transplantation that preserves spontaneous breathing function — This intervention uses a spontaneous-breathing-preserving anesthesia strategy during lung transplantation, which differs from conventional management based on endotracheal intubation and invasive mechanical ventilation. A supraglottic airway (laryngeal mask airway) is used when feasible instead of endotracheal intubation to maintain spontaneous breathing throughout the procedure. Neuromuscular blocking agents are minimized, and regional nerve blocks (such as intercostal nerve blocks or paravertebral blocks) are used to control pain and suppress cough while preserving the patient's ability to breathe independently. After surgery, patients receive protocol-guided noninvasive respiratory support (for example, high-flow nasal oxygen or noninvasive ventilation), with the goal of avoiding routine invasive mechanical ventilation.

SUMMARY:
The goal of this prospective, multicenter, single-arm clinical study is to learn whether a breathing-preserved anesthesia-surgical strategy can improve early recovery and perioperative survival in adults undergoing rescue/bridge lung transplantation.

The main questions it aims to answer are whether, in adult rescue lung transplant recipients, a breathing-preserved anesthesia-surgical strategy can improve early postoperative recovery and perioperative survival, with a focus on the need for postoperative invasive mechanical ventilation, postoperative length of hospital stay, and perioperative survival outcomes.

Participants will undergo lung transplantation using a standardized breathing-preserved anesthesia-surgical pathway, with predefined criteria for conversion to endotracheal intubation and/or initiation or escalation of extracorporeal support when clinically necessary. Participants will receive standardized perioperative care per each participating center's transplant pathways and will be followed from screening through hospital discharge and up to 30 days after surgery. Routine perioperative data and key postoperative outcomes, including major complications (e.g., graft dysfunction, respiratory support events, infections, bleeding requiring re-intervention, acute kidney injury, rejection, and thrombotic events), will be collected.

DETAILED DESCRIPTION:
Purpose:

Rescue/bridge lung transplantation recipients represent a high-risk population with limited physiologic reserve and a high likelihood of prolonged postoperative support. This prospective, multicenter, single-arm clinical study (BREATH-Rescue) aims to evaluate the clinical effectiveness and perioperative safety of a breathing-preserved anesthesia-surgical strategy designed to minimize exposure to invasive mechanical ventilation while maintaining adequate gas exchange and hemodynamic stability. The study focuses on early postoperative recovery and perioperative survival, with primary outcomes centered on postoperative invasive mechanical ventilation (IMV) requirement, postoperative hospital length of stay (LOS), and perioperative survival through hospital discharge or 30 days after surgery (whichever occurs first).

Study Design and Methods:

BREATH-Rescue will enroll approximately 40 adult (≥18 years) rescue/bridge lung transplant candidates across multiple centers, with an anticipated ~36 participants contributing evaluable data for primary endpoint analyses. Rescue/bridge status is defined by meeting any of the following conditions prior to transplantation: ongoing invasive mechanical ventilation (endotracheal tube or tracheostomy), receipt of ECMO/other extracorporeal life support (ECLS), or urgent escalation of support due to progressive respiratory and/or circulatory failure prompting an emergency transplant pathway. Key baseline organ function thresholds are applied (e.g., LVEF ≥40%, eGFR ≥40 mL/min/1.73 m²), with exclusion of active uncontrolled infection.

All participants will undergo lung transplantation under a standardized breathing-preserved anesthesia-surgical pathway. The strategy emphasizes preservation or early restoration of spontaneous breathing when feasible, use of a laryngeal mask airway-based approach and intravenous anesthesia with multimodal analgesia/regional techniques, and continuous physiologic monitoring. Predefined criteria guide prompt conversion to endotracheal intubation and/or initiation or escalation of extracorporeal support when clinically necessary (e.g., inadequate oxygenation/ventilation, severe hypercapnia/acidosis, hemodynamic instability, major airway bleeding, insufficient operative exposure, or airway device failure). Postoperatively, participants will receive standardized perioperative management per center transplant pathways. Outcomes and safety events will be collected from screening through hospital discharge and up to 30 days after surgery, including key complications (e.g., primary graft dysfunction graded at 0/24/48/72 hours, respiratory support events such as re-intubation/tracheostomy/new or escalated ECMO, infections, bleeding requiring re-intervention, acute kidney injury, rejection episodes, and thrombotic events). The primary endpoint is a composite of three early recovery metrics (reported both as a composite and as individual components): postoperative IMV requirement, postoperative LOS, and perioperative survival.

Anticipated Results:

Investigators hypothesize that, in rescue/bridge lung transplant recipients, implementation of a breathing-preserved anesthesia-surgical strategy will increase the proportion of patients who do not require postoperative IMV, shorten postoperative hospital LOS, and achieve an acceptable perioperative survival rate through discharge or 30 days, compared with participating centers' historical outcomes under conventional intubated strategies. The study is expected to generate pragmatic, multicenter evidence on feasibility, safety signals (including conversion/intubation and ECMO escalation rates), and recovery trajectories in this high-risk population, thereby informing pathway standardization and the design of future controlled comparative studies.

ELIGIBILITY:
[1] Inclusion Criteria

1. Age and informed consent: Age ≥18 years. The participant or their legally authorized representative (LAR) is able to complete the informed consent process in a rescue/emergent transplant setting and sign written informed consent.
2. Transplant candidacy: Listed in the China Lung Transplantation Registry (CLuTR) or the lung transplant waiting list of the participating center, with a planned allogeneic lung transplantation.
3. Rescue/bridge definition (core cohort criterion): Meets any of the following conditions and is deemed by the study team to require rescue/emergent transplantation and to proceed to transplant: continuous invasive mechanical ventilation preoperatively (endotracheal intubation or tracheostomy); or preoperative extracorporeal membrane oxygenation (ECMO) / other extracorporeal life support (ECLS); or urgent escalation of support due to progressive respiratory and/or circulatory failure, entering a rescue transplant pathway.
4. Minimum key organ function: Left ventricular ejection fraction (LVEF) ≥40%; estimated glomerular filtration rate (eGFR) ≥40 mL/min/1.73 m²; no evidence of acute liver failure or decompensated cirrhosis/portal hypertension; American Society of Anesthesiologists (ASA) Physical Status classification ≤ IV.
5. Infection and transmissible diseases: No evidence of active infection; no active tuberculosis; HIV/HBV/HCV meet the center's transplant requirements (e.g., undetectable viral load, as applicable).
6. Rehabilitation and support: Demonstrated potential for postoperative rehabilitation (able to cooperate with training) and reliable caregiving support (at least one primary caregiver).

[2] Exclusion Criteria

1. Informed consent/adherence: Refusal of or withdrawal of informed consent; investigator judgment that follow-up cannot be completed or that there is repeated serious non-adherence.
2. Transplant type: Re-transplantation, multi-organ transplantation, or planned lobar lung transplantation.
3. Recent major cardiovascular/cerebrovascular events: Acute coronary syndrome/myocardial infarction or stroke within the past 30 days.
4. Severe organ dysfunction/acute failure: LVEF <40%; eGFR <40 mL/min/1.73 m²; acute liver failure or decompensated cirrhosis/portal hypertension; acute renal failure requiring dialysis with low likelihood of recovery; significant preoperative neuropsychiatric disorder or impaired consciousness.
5. High risk of severe infection: Septic shock; active extrapulmonary/disseminated infection; active tuberculosis; detectable HIV viral load (or otherwise not meeting the center's transplant criteria).
6. High risk of major bleeding: Severe bronchiectasis not treated with preoperative vascular intervention or not readily correctable.
7. Malignancy: Active malignancy or malignancy with high risk of recurrence or cancer-related mortality.
8. Severe chest wall or spinal deformity: Deemed by the study team to compromise surgical exposure, ventilation/airway management, or perioperative safety.
9. Substance use/dependence: Current smoking, e-cigarette/vaping use, inhaled cannabis use, or intravenous drug use.
10. Tubeless/breathing-preserved strategy not safely feasible: The anesthesia team judges a difficult airway or laryngeal mask/non-intubated airway management to be unsafe (e.g., anticipated difficult airway, pharyngeal/laryngeal stenosis unsuitable for laryngeal mask, or other conditions unfavorable for airway management), including but not limited to: Mallampati class >III, mouth opening <3 cm, thyromental distance <5 cm, or significant airway anatomical variation (e.g., anomalous right upper lobe bronchial origin in a planned right lung transplantation) such that safe management with a laryngeal mask or single-lumen tube is deemed unlikely.
11. Donor/donor lung limitations: Donor age >60 years; donor mechanical ventilation >14 days; positive donor airway microbiology that the transplant team deems unacceptable.
12. Protected population: Pregnant or breastfeeding women.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Requiring Postoperative Invasive Mechanical Ventilation (IMV) During Index Hospitalization | From ICU admission immediately after leaving the operating room until hospital discharge or in-hospital death, assessed up to 90 days postoperatively (if hospitalization extends beyond 90 days, events after day 90 will not be counted for this outcome).
  Number of participants who require postoperative invasive mechanical ventilation (IMV) delivered via an endotracheal tube or tracheostomy tube at any time after leaving the operating room and before hospital discharge (including in-hospital death).
  Time Frame: From post-anesthesia care/ICU admission (immediately after leaving the operating room) through hospital discharge or in-hospital death (index hospitalization)
Postoperative Hospital Length of Stay (Days) During Index Hospitalization | From end of surgery (postoperative Day 0) until hospital discharge or in-hospital death (index hospitalization), assessed up to 90 days.
  The number of days from the end of surgery (postoperative Day 0) to the date the participant is discharged from the index hospitalization, according to institutional discharge criteria. Participants who die in hospital will be assigned length of stay through the date of in-hospital death.
Rate of Perioperative Survival | From start of transplant surgery through hospital discharge or postoperative Day 30, whichever occurs first.
  Perioperative survival is defined as the proportion of participants who remain alive from the start of transplant surgery through hospital discharge or postoperative Day 30, whichever occurs first. Participants who die before discharge or before postoperative Day 30 will be counted as non-survivors for this outcome.

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data (IPD) underlying the analyses of this clinical study, limited to baseline and perioperative variables. Baseline IPD will include demographics (e.g., age, sex), primary diagnosis, key comorbidities, and transplant-relevant preoperative measures and donor/recipient characteristics recorded in structured fields. Perioperative IPD will include operative and anesthesia strategy, airway management, intraoperative/early postoperative respiratory and hemodynamic parameters, major perioperative interventions (e.g., ECMO use), and key in-hospital outcomes during the index hospitalization (e.g., need for postoperative IMV, complications, ICU/hospital length of stay, and in-hospital mortality). The study protocol and statistical analysis plan will also be shared. All direct identifiers will be removed and dates will be shifted/aggregated as needed to protect privacy.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning at study completion and ending 2 years after study completion.
Access Criteria: De-identified IPD and supporting documents (study protocol, statistical analysis plan, and data dictionary) will be available to qualified researchers outside the primary study group for scientifically sound research purposes. Access will be granted upon submission of a written request that includes a brief research proposal, analysis plan, and proof of relevant ethics/IRB review if applicable. Requests will be reviewed by the study steering committee/data access committee. Approved requestors must sign a data use agreement prohibiting re-identification attempts and onward sharing, and requiring appropriate data security measures and acknowledgement of the original study. Data will be provided through a secure electronic transfer or a controlled-access online repository; access instructions will be provided after approval.
URL: https://www.gyfyyy.cn/